CLINICAL TRIAL: NCT06846554
Title: A Phase 2, Multicentre, Open-Label Trial to Evaluate APL-9796 in Adult Participants With Pulmonary Hypertension (ViTAL-PH)
Brief Title: A Trial of "APL-9796'' in Adults With Pulmonary Hypertension
Acronym: ViTAL-PH
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Apollo Therapeutics Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AP13CP02
Record Dates: First submitted 2025-01-10; First posted 2025-02-26 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary Hypertension; WHO group 3; WHO group 1 PH
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension, Pulmonary

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part A: in adults with WHO Group 1 PAH. (Experimental): Three (3) APL-9796 dose levels are planned for evaluation using BOIN design.
  Interventions: Drug: APL-9796
- Part B (optional): in adults with WHO Group 3 PH-ILD (Experimental): Cohorts will be enrolled sequentially at N=4, at a dose level determined by the Safety Review Committee (SRC) based on data from Part A.
  Interventions: Drug: APL-9796

INTERVENTIONS:
Drug: APL-9796 — 3 Cohorts are planned in Part A.
  Arms: Part A: in adults with WHO Group 1 PAH.
Drug: APL-9796 — The decision to initiate optional Part B in WHO Group 3 PH-ILD participants will be made by the Safety Review Committee (SRC).
  Arms: Part B (optional): in adults with WHO Group 3 PH-ILD

SUMMARY:
The AP13CP02 study is a phase 2, open-label, dose escalation trial to determine how safe and tolerable multiple subcutaneous (SC) injections of APL-9796 are for patients with PH. The study will also assess how effective APL-9796 could be for treating patients with PH and whether the body produces antibodies working against APL-9796.

The trial will be conducted in two parts:

* Part A: Up to 36 adults with WHO Group 1 Pulmonary arterial hypertension (PAH).
* Part B (optional): Up to 12 adults with WHO Group 3 - PH associated with ILD (PH-ILD).

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be 18 to 80 years of age inclusive
2. Participants who are diagnosed with pulmonary hypertension via right heart catheterisation (RHC), documented at any time prior to Screening.
3. WHO Functional Class II or III
4. Participant has the CardioMEMS PA Sensor implanted.

Exclusion Criteria:

1. Hospital admission related to PH within 3 months prior to Screening.
2. Major surgical procedure within 3 months prior to Screening, unless participant is assessed as completely recovered by the Investigator
3. Diagnosis of PH due to human immunodeficiency virus, portal hypertension, schistosomiasis, or uncorrected congenital heart disease
4. History of left-sided heart disease and/or clinically significant cardiac disease
5. History of uncontrolled systemic hypertension
6. eGFR ≤30 ml/min/1.73m2
7. Life expectancy of < 12 months, as assessed by the Investigator
8. Diagnosed with a malignancy within 5 years of enrolment
9. Contraindications to protocol-required imaging (MRI), diagnostic, or sampling methods

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-04-09 (Actual); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Through study completion (approximately 2 years)
  Number of participants who experience Treatment-Emergent Adverse Events will be reported which also include the frequency, severity (CTCAE V5.0) and relationship (causality) of AEs

SECONDARY OUTCOMES:
To assess the Telemetry Parameters | from baseline (CFB) to Day 169
  Telemetry parameter is assessed using Total pulmonary resistance (TPR)
To assess the Telemetry Parameters | from baseline (CFB) to Day 169
  Telemetry parameter is assessed using Pulmonary arterial pressures: systolic, diastolic and mean (mPAP)
To assess Six minute walk test / Six minute walk distance (6MWD) | from baseline (CFB) to Day 169
  A 6-minute walk test (6MWT) is assessed per the guidelines of the American Thoracic Society 2003
To assess NT-proB-type Natriuretic Peptide (NT-proBNP) | from baseline (CFB) to Day 169
  The level of NT-proBNP is assessed by blood sample collection and analysis
To assess the Quality of life | from baseline (CFB) to Day 169
  Quality of life is assessed using SF-36 questionnaire
To assess the Quality of life | from baseline (CFB) to Day 169
  Quality of life is assessed using emPHasis-10 questionnaire
To evaluate the PK of APL-9796 in participants with PH | at each visit (approximately every 28 days until day 169), then day 254, day 339 and day 508
  APL-9796 concentrations in serum
To evaluate the immunogenicity of APL-9796 in participants with PH. | at each visit (approximately every 28 days until day 169), then day 254, day 339 and day 508
  * Incidence of anti-drug antibody (ADA) against APL-9796 (including titres)
  * Incidence of neutralising antibody (Nab) against APL-9796 (including titres)

CONTACTS AND LOCATIONS:
Locations (4):
- United Kingdom (4):
  - Hammersmith/Imperial Hospital, London, London
  - Royal United Hospital Bath, Bath
  - Royal Brompton Hospital, London
  - Sheffield Teaching Hospitals, Sheffield